CLINICAL TRIAL: NCT04759586
Title: A Randomized Phase 3 Trial of Nivolumab (NSC# 748726) in Combination With Chemo-Immunotherapy for the Treatment of Newly Diagnosed Primary Mediastinal B-Cell Lymphoma
Brief Title: Nivolumab in Combination With Chemo-Immunotherapy for the Treatment of Newly Diagnosed Primary Mediastinal B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-01071; NCI-2021-01071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANHL1931 (Other: Children's Oncology Group); ANHL1931 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Primary Mediastinal Large B-Cell Lymphoma
MeSH Terms: interventions — Specimen Handling; Biopsy; Cyclophosphamide; Doxorubicin; etoposide phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Spinal Puncture; Nivolumab; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Magnetic Resonance Spectroscopy; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Rituximab; CT-P10; Hyaluronoglucosaminidase; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (DA-EPOCH-R) (Active Comparator): See Detailed Description
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Biological: Filgrastim; Procedure: Lumbar Puncture; Biological: Pegfilgrastim; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Vincristine Sulfate
- Arm B (DA-EPOCH-R, nivolumab) (Experimental): Patients receive treatment as in Arm A. Patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO and LP for CSF collection during screening. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Biological: Filgrastim; Procedure: Lumbar Puncture; Biological: Nivolumab; Biological: Pegfilgrastim; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Vincristine Sulfate
- Arm C (R-CHOP) (Active Comparator): Patients receive prednisone or prednisolone PO QD on days 1-5 and rituximab IV or rituximab and hyaluronidase human SC over 5 minutes on day 1 or 5. Patients also receive cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV over 1-15 minutes or up to 60 minutes, and vincristine sulfate IV over 1 or up to 60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Vincristine Sulfate
- Arm D (R-CHOP, nivolumab) (Experimental): Patients receive treatment as in Arm C. Patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Biological: Nivolumab; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Vincristine Sulfate
- Arm E (R-CHOP, radiation therapy) (Active Comparator): Patients receive treatment as in Arm C. Within 6-8 weeks after completion of chemotherapy, patients undergo radiation therapy over 25 fractions. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Radiation: Radiation Therapy; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Vincristine Sulfate
- Arm F (R-CHOP, nivolumab, radiation therapy) (Experimental): Patients receive treatment as in Arm D. Within 6-8 weeks after completion of chemotherapy, patients undergo radiation therapy over 25 fractions. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Biological: Nivolumab; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Radiation: Radiation Therapy; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
  Arms: Arm A (DA-EPOCH-R); Arm B (DA-EPOCH-R, nivolumab)
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
  Arms: Arm A (DA-EPOCH-R); Arm B (DA-EPOCH-R, nivolumab)
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm B (DA-EPOCH-R, nivolumab); Arm D (R-CHOP, nivolumab); Arm F (R-CHOP, nivolumab, radiation therapy)
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
  Arms: Arm A (DA-EPOCH-R); Arm B (DA-EPOCH-R, nivolumab)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisolone — Given PO
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm E (R-CHOP, radiation therapy); Arm F (R-CHOP, nivolumab, radiation therapy)
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm A (DA-EPOCH-R); Arm B (DA-EPOCH-R, nivolumab); Arm C (R-CHOP); Arm D (R-CHOP, nivolumab); Arm E (R-CHOP, radiation therapy)

SUMMARY:
This phase III trial compares the effects of nivolumab with chemo-immunotherapy versus chemo-immunotherapy alone in treating patients with newly diagnosed primary mediastinal B-cell lymphoma (PMBCL). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Treatment for PMBCL involves chemotherapy combined with an immunotherapy called rituximab. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving nivolumab with chemo-immunotherapy may help treat patients with PMBCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if nivolumab + chemo-immunotherapy results in a superior long term progression-free survival (PFS) (events defined as disease progression confirmed by central review or death) when compared with chemo-immunotherapy alone in patients with newly diagnosed primary mediastinal B-cell lymphoma.

SECONDARY OBJECTIVES:

I. To compare the rates of "efficacy-related event-free survival (EFS)" (eEFS) (events defined as progression, change in therapy due to finding that led to concern about efficacy, biopsy + disease after 6 cycles of therapy, or death) between chemo-immunotherapy alone and chemo-immunotherapy + nivolumab in patients with newly diagnosed PMBCL.

II. To compare the rates of "therapy-related EFS" (tEFS) (events defined as relapse/progression, change in therapy for any reason, biopsy + disease after 6 cycles of therapy, secondary malignancy [SMN] or death) between chemo-immunotherapy alone and chemo-immunotherapy + nivolumab in patients with newly diagnosed PMBCL.

III. To compare the rates of overall survival (OS) between chemo-immunotherapy alone and chemo-immunotherapy + nivolumab in patients with newly diagnosed PMBCL.

IV. To establish the rate of a positive positron emission tomography (PET)-computed tomography (CT) (defined as Deauville score 4 or 5) at the completion of 6 cycles of nivolumab + rituximab (R)- cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP)/dose-adjusted (DA)-etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (EPOCH)-R and R-CHOP/DA-EPOCH-R in patients with newly diagnosed PMBCL and evaluate the prognostic significance of such a finding.

EXPLORATORY OBJECTIVES:

I. To bank radiology images for further studies. II. To bank specimens for future correlative studies. III. Characterize the immune profile of patients treated with nivolumab + chemo-immunotherapy to identify markers predictive of response.

IV. Define the rate of complete response at the completion of initial planned therapy.

OUTLINE: Patients are randomly assigned to backbone therapy or backbone therapy + nivolumab within each of 6 strata. The strata are determined by physician's choice of backbone (DA-EPOCH-R versus [vs.] R-CHOP vs. R-CHOP + RT) and whether or not the patient had 1 prior cycle of therapy.

ARM A (DA-EPOCH-R): Patients receive prednisone or prednisolone orally (PO) once daily (QD) on days 1-5 and rituximab intravenously (IV) or rituximab and hyaluronidase human subcutaneously (SC) over 5 minutes on day 1 or 5. Patients also receive etoposide phosphate, doxorubicin hydrochloride, and vincristine sulfate IV over 96 hours on days 1-4 and cyclophosphamide IV over 30-60 minutes on day 5. Beginning 24-72 hours after completing cyclophosphamide, patients receive filgrastim or pegylated filgrastim SC daily until absolute neutrophil count (ANC) is >= 500/uL after the expected nadir. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) during screening and as clinically indicated and a lumbar puncture (LP) for cerebral spinal fluid (CSF) collection optionally during screening. Patients also undergo computed tomography (CT) or positron emission tomography (PET)/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

ARM B (DA-EPOCH-R + NIVOLUMAB): Patients receive treatment as in Arm A. Patients also receive nivolumab IV over 30 minutes on day 1. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

ARM C (R-CHOP): Patients receive prednisone or prednisolone PO QD on days 1-5 and rituximab IV or rituximab and hyaluronidase human SC over 5 minutes on day 1 or 5. Patients also receive cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV over 1-15 minutes or up to 60 minutes, and vincristine sulfate IV over 1 or up to 60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

ARM D (R-CHOP + NIVOLUMAB): Patients receive treatment as in Arm C. Patients also receive nivolumab IV over 30 minutes on day 1. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

ARM E (R-CHOP + RADIOTHERAPY): Patients receive treatment as in Arm C. Within 6-8 weeks after completion of chemotherapy, patients undergo radiation therapy over 25 fractions. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

ARM F (R-CHOP + RADIOTHERAPY + NIVOLUMAB): Patients receive treatment as in Arm D. Within 6-8 weeks after completion of chemotherapy, patients undergo radiation therapy over 25 fractions. Patients undergo ECHO during screening and as clinically indicated and LP for CSF collection optionally during screening. Patients also undergo CT or PET/CT throughout the trial. Additionally, patients undergo bone marrow biopsy and aspiration optionally during screening and as clinically indicated on study. Patients undergo blood sample collection on study.

After completion of study treatment, patients are followed up every 3 months for year 1, every 6 months for years 2-3, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 2 years
* Patient must have histologically confirmed primary mediastinal B-cell lymphoma (PMBCL) as defined by World Health Organization (WHO) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 or ECOG performance status of 3 if poor performance is related to lymphoma

  * Children's Oncology Group (COG) Institutions: Use Karnofsky for patients >= 17 and < 18 years of age and Lansky for patients < 17 years of age
* Adults (age 18 or older): Creatinine clearance >= 30 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within 28 days prior to registration. Estimated creatinine clearance is based on actual body weight
* Pediatric Patients (age < 18 years): The following must have been obtained within 14 days prior to registration:

  * Measured or calculated (based on institutional standard) creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2, or
  * Serum creatinine =< 1.5 x institutional upper limit of normal (IULN), or a serum creatinine based on age/sex as follows:

    * Age : 2 to < 6 year; Maximum serum creatinine (mg/dL): 0.8 (male; 0.8 (female)
    * Age : 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 (male); 1 (female)
    * Age : 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
    * Age : 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
    * Age : >= 16 years to < 18 years; Maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* Patients with abnormal liver function will be eligible to enroll if the lab abnormality is thought to be due to the lymphoma or Gilbert's syndrome
* Age >= 18 years: Ejection fraction of >= 50% by echocardiogram
* Age < 18 years: Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by radionuclide angiogram
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Administration of prior anti-cancer therapy except as outlined below:

  * A short course (=< 2 weeks) of corticosteroids for the relief of lymphoma-related symptoms
  * A single course of COP (cyclophosphamide, vincristine, and prednisone)
  * One cycle of chemo-immunotherapy including R-CHOP, DA-EPOCH-R, a pediatric mature B-cell non-Hodgkin lymphoma (B-NHL) induction therapy (such as ANHL1131), or intrathecal chemotherapy that has not started more than 21 days prior to enrollment
* Active ischemic heart disease or heart failure
* Active uncontrolled infection
* Central nervous system (CNS) involvement of lymphoma
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of this trial
* Active autoimmune disease that has required systemic treatment (such as disease modifying agents, corticosteroids, or immunosuppressive agents) in the past 2 years. Replacement therapy such as thyroxine, insulin or physiologic corticosteroid for adrenal or pituitary insufficiency is not considered a form of systemic treatment
* In patients < 18 years of age hepatitis B serologies consistent with past or current infections
* Patients with severe hepatic impairment (Child-Pugh class C or serum total bilirubin > 5.0 mg/dL) unless thought to be due to lymphoma or Gilbert's syndrome
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Sexually active patients of reproductive potential who have not agreed to use a highly effective contraceptive method (failure rate of < 1% per year when used consistently and correctly) for the duration of their study participation
* Lactating females are not eligible unless they have agreed not to breastfeed their infants starting with the first dose of study therapy and for at least 6 months after the last dose of rituximab

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From enrollment on the study to first occurrence of relapse/progression or death, assessed up to 7 years
  The primary analysis will be a one-sided Log-rank test stratified by choice of backbone and radiation therapy and whether the patient had a cycle of therapy prior to enrolling.

SECONDARY OUTCOMES:
Efficacy-related event-free survival | Up to 7 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as progression, change in therapy due to a finding that led to concern about efficacy, biopsy + disease after 6 cycles of therapy, and death.
Therapy-related event-free survival | Up to 7 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as progression, change in therapy due to a finding that led to concern about efficacy, biopsy + disease after 6 cycles of therapy, and death.
Overall survival | Up to 7 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as only death.
Proportion of positive positron emission tomography (PET) scans | Up to 6 cycle (1 cycle = 21 days)
  Will be analyzed descriptively with a point estimate and Clopper-Pearson 95% confidence interval in the trial overall and in each treatment arm separately. The prognostic significance of positive PET after 6 cycles of therapy will be evaluated using a Cox proportional hazards regression on PFS with PET result (positive versus [vs.] negative), choice of backbone (rituximab [R]-cyclophosphamide, doxorubicin, vincristine, and prednisone [CHOP] + radiation therapy [RT] regardless of end-of-therapy imaging vs. R-CHOP without RT unless biopsy positive at end-of-therapy vs. dose-adjusted [DA]-etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin [EPOCH]-R without RT unless biopsy positive at end of therapy), and assignment to nivolumab (yes vs. no) as covariates.

OTHER OUTCOMES:
Immune profile of patients treated with nivolumab + chemo-immunotherapy | Up to 7 years
  Analysis will be by paired t-test (for pre- vs. post-treatment measurements) or two-sample equal-variance t-test (for comparisons of nivolumab vs. non-nivolumab or responders [complete response/partial response] vs. non-responders [stable disease/progressive disease]).
Complete response rate | At the completion of initial planned therapy
  Will be described using point estimates and Clopper-Pearson 95% confidence intervals for the complete response rate overall and in each treatment arm separately.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Roth, Principal Investigator — Children's Oncology Group
Locations (233):
- United States (215):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - New York Medical College, Valhalla, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
- Australia (5):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm